CLINICAL TRIAL: NCT05818449
Title: Improvement of Personalized Cancer Care for Patients With Advanced Non-Small Cell Lung Cancer (NSCLC) Through Digital Connection of Specialized Cancer Centers, Community Hospitals, Private Practices and Patients (DigiNet)
Brief Title: Improvement of Personalized Lung Cancer Care Through Digital Connection and Patient Participation (DigiNet)
Acronym: DigiNet
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cologne (Other)
Collaborators: Gemeinsamer Bundesausschuss (G-BA) (Unknown); AOK Rheinland/Hamburg (Industry); AOK Nordwest (Industry); BARMER (Other); University Hospital, Essen (Other); Charite University, Berlin, Germany (Other); Berlin Institute of Health (Other); Helios Klinikum Emil von Behring (Unknown); University Hospital Carl Gustav Carus (Other); Deutsche Krebsgesellschaft e.V. (Other); Berufsverband der Niedergelassenen Hämatologen und Onkologen in Deutschland e.V. (Unknown); AOK Bundesverband (Unknown); FOM Hochschule für Oekonomie und Management (Unknown); University Medicine Greifswald (Other); Technische Universität Dresden (Other)
Responsible Party: Principal Investigator, Prof. Dr. Juergen Wolf, Prof. Dr., University of Cologne
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01NVF20021
Record Dates: First submitted 2022-12-12; First posted 2023-04-18 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Non-small Cell Lung Cancer Stage IV
Keywords: Carcinoma, Non-Small-Cell Lung; Carcinoma, Non-Small-Cell Lung* / diagnosis; Carcinoma, Non-Small-Cell Lung* / genetics; Precision Medicine; Pathology, Molecular; Patient Reported Outcome Measures; Database Management Systems
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Carcinoma; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DigiNet group (Experimental): The intervention group will receive the DigiNet intervention.
  Interventions: Other: DigiNet intervention
- Comparison group (No Intervention): The comparison group will receive usual care.

INTERVENTIONS:
Other: DigiNet intervention — Patients with initial diagnosis of NSCLC stage IV in the model region receiving the following interventions:
  * broad NGS-based molecular diagnostics and, based thereupon, personalized treatment information within the national Network Genomic Medicine (nNGM) lung cancer
  * regular clinical follow-up visits and data documentation in the shared central digital database by participating physicians
  * monthly assessment of patient-reported outcomes (PRO) on quality of life, anxiety, and depression
  * incorporation of PROs into treatment by physicians
  * treatment monitoring and counseling in the case of critical conditions by expert committee
  Arms: DigiNet group

SUMMARY:
The aim of the DigiNet project is to improve the treatment of patients with advanced non-small cell lung cancer (NSCLC) in Germany. The project promotes the transfer of the latest scientific knowledge into standard care. The DigiNet project is based on the established precision medicine program, the National Network Genomic Medicine Lung Cancer (nNGM) in Germany, whereby every patient receives molecular diagnostics and personalized therapy information after the initial diagnosis. Within the framework of the DigiNet project, specialized academic centers will be digitally connected with practitioners via a shared project database. Furthermore, a committee of experts will monitor the course of treatment and will advise the practitioners in case of critical conditions. Additionally, patient-reported outcomes will be incorporated into the treatment.

DETAILED DESCRIPTION:
The aim of the DigiNet project is to prospectively evaluate a precision medicine program for lung cancer and to improve personalized care of patients with advanced non-small cell lung cancer (NSCLC) through a collaboration of specialized academic centers with routine care providers (hospitals, oncology practices). The use of targeted therapies will be regularly monitored and guided through a shared digital database. Patients with an initial diagnosis of stage IV NSCLC in the study regions (study region east: Berlin and Saxony; study region west: North Rhine-Westphalia) are included. DigiNet builds on the foundations and structures of the National Network Genomic Medicine Lung Cancer (nNGM) in Germany, which provides molecular diagnostics and treatment information to the participating physicians based on the latest evidence.

Within the framework of DigiNet, patients are regularly consulted by the study practitioners and the clinical data is documented in a structured manner in a central project database. Through the digital collaboration of the nNGM network centers via the shared project database with the practitioners in routine care, continuous monitoring of the course of treatment and, in the case of critical conditions, treatment guidance by an expert committee advising the practitioner is provided. In addition, the patients routinely assess the quality of life (EORTC QLQ-C30, EORTC QLQ-LC29, EQ-5D), as well as anxiety and depression (PHQ-4). The results of these patient-reported outcomes (PROs) are incorporated into the treatment by the practitioners (patient-centered treatment approach).

The evaluation of the project is structured into different core domains: An evaluation of clinical endpoints, process parameters (implementation of the intervention), and health economic evaluations will be conducted. The acceptance and potential for improvement of the project will be assessed through qualitative interviews with the stakeholders. Data from the state cancer registries of the study regions will be incorporated to generate a population-based comparative cohort for the evaluation of the main research questions of DigiNet, thereby representing patients receiving routine care in Germany.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with advanced NSCLC, stage IV
* Age > 18 years
* Life expectancy at least 4 weeks (initial assessment at inclusion in nNGM and confirmation at baseline (implementation of treatment decision))

Exclusion Criteria:

* Missing informed consent
* Illnesses and behaviors that impair compliance (e.g., dementia, addictive disorders)
* Severely impaired general physical condition that no longer permits therapy for lung cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 850 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | up to 34 months
  Overall Survival (OS) will be assessed in months.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | up to 34 months
  Progression-Free Survival (PFS) will be assessed in months.
Time on First Treatment (ToT) | up to 34 months
  Duration under first-line therapy will be assessed in months.
Hospitalization rate | up to 34 months
  Frequency of hospital stays will be assessed using health insurance data.
Quality of Life (EORTC QLQ-C30) | up to 34 months
  Quality of Life (European Organisation for Research and Treatment of Cancer, Quality of Life Core Questionnaire, EORTC QLQ-C30) will be assessed in absolute values and change over time. Each item is rated on a response scale 1 = "not at all" to 4 = "very much" with exception of the last two items, which assess overall health and quality of life on a scale from 1 = "very poor" to 7 = "excellent". All EORTC QLQ-C30 scale scores range from 0 to 100, whereby higher scores on a functional scale indicate a high level of functioning, whereas higher scores on a symptom scale/symptom item indicate greater symptom burden.
Quality of Life (EORTC QLQ-LC29) | up to 34 months
  Quality of Life (European Organisation for Research and Treatment of Cancer, Quality of Life Questionnaire Lung Cancer, EORTC QLQ-LC29) will be assessed in absolute values and change over time. Each item is rated on a response scale 1 = "not at all" to 4 = "very much" and refer to the time frame "during the past week". All EORTC QLQ-LC29 scale scores range from 0 to 100, whereby higher scores for a symptom scale/symptom item indicate greater symptom burden.
Symptoms of anxiety (GAD-2) | up to 34 months
  Symptoms of anxiety (Generalized Anxiety Disorder Scale-2, GAD-2) will be assessed in absolute values and change over time. Each item is rated on a response scale 0 = "not at all" to 3 = "nearly every day" and refer to the time frame "during the past two weeks". Higher scores indicate greater symptom burden.
Symptoms of depression (PHQ-2) | up to 34 months
  Symptoms of depression (Patient-Health-Questionnaire-2, PHQ-2) will be assessed in absolute values and change over time. Each item is rated on a response scale 0 = "not at all" to 3 = "nearly every day" and refer to the time frame "during the past two weeks". Higher scores indicate greater symptom burden.
Frequency of applied targeted molecular therapies based on clinical therapy information from the MURIEL database | up to 34 months
  The frequency of applied targeted molecular therapies is based on clinical therapy information from the MURIEL database.
Frequency of active contact of the expert advisory board with physicians during the course of treatment | up to 34 months
  Assessing the frequency of the expert advisory board actively contacting physicians during the course of treatment
Completeness of the documentation of the treatment course | up to 34 months
  Assessing the completeness of the documentation of the treatment course (DigiNet study visits) in %.
Frequency of patients' completing the PROs | up to 34 months
  Assessing the frequency of patients' completing the patient-reported outcomes (PRO) via the internet portal
Cost-effectiveness of DigiNet compared to standard care in terms of incremental costs per life years gained | up to 34 months
  Assessing the cost-effectiveness of DigiNet compared to standard care in terms of incremental costs per life years gained
Cost-effectiveness of DigiNet compared to standard care in terms of costs per quality-adjusted life year [QALY] | up to 34 months
  Assessing the cost-effectiveness of DigiNet compared to standard care in terms of costs per quality-adjusted life year [QALY]
Cost of implementation related to DigiNet from the service provider perspective (hospital, practices) | up to 34 months
  Assessing the cost of implementation related to DigiNet from the service provider perspective (hospital, practices) in Euro (€)
Process costs related to DigiNet from the service provider perspective (hospital, practices) | up to 34 months
  Assessing the process costs related to DigiNet from the service provider perspective (hospital, practices) in Euro (€)
Formative evaluation | up to 34 months
  Formative evaluation regarding the implementation will be conducted using qualitative analysis of semi-structured interviews

CONTACTS AND LOCATIONS:
Overall Officials: Jürgen Wolf, Prof. Dr., Principal Investigator — Uniklinik Köln
Locations (41):
- Germany (41):
  - Universitätsklinikum Würzburg, Würzburg, Bavaria
  - Hämatologisch-Onkologische Schwerpunktpraxis, Bad Liebenwerda, Brandenburg
  - Universitätsklinikum Aachen, Aachen, North Rhine-Westphalia
  - Johanniter-Krankenhaus Bonn, Bonn, North Rhine-Westphalia
  - Onkozentrum Bonn, Bonn, North Rhine-Westphalia
  - Universitätsklinikum Bonn (UKB), Bonn, North Rhine-Westphalia
  - Zentrum für ambulante Hämatologie und Onkologie Rhein-Sieg (ZAHO), Brühl, North Rhine-Westphalia
  - MV-Zentrum für Hämatologie und Onkologie, Cologne, North Rhine-Westphalia
  - Universitätsklinikum Köln, Cologne, North Rhine-Westphalia
  - MVZ West GmbH Standort Köln-Kalk, Cologne, North Rhine-Westphalia
  - Praxis Internistischer Onkologie und Hämatologie (pioh), Cologne, North Rhine-Westphalia
  - Gemeinschaftspraxis für Hämatologie & Onkologie, Dortmund, North Rhine-Westphalia
  - Universitätsklinikum Essen, Essen, North Rhine-Westphalia
  - Praxis für Hämatologie und Internistische Onkologie, Hamm, North Rhine-Westphalia
  - Klinikum Leverkusen, Leverkusen, North Rhine-Westphalia
  - Kliniken Maria Hilf GmbH, Mönchengladbach, North Rhine-Westphalia
  - MVZ für Hämatologie und Onkologie, Mülheim, North Rhine-Westphalia
  - Praxis und Tagesklinik für Internistische Onkologie und Hämatologie, Recklinghausen, North Rhine-Westphalia
  - Krankenhaus Bethanien Solingen, Solingen, North Rhine-Westphalia
  - Onkologie Rheinsieg, Troisdorf/Bonn-Beuel/Bad Honnef, North Rhine-Westphalia
  - MVZ Medizinisches Versorgungszentrum am Marien-Hospital Wesel, Wesel, North Rhine-Westphalia
  - Medizinisches Versorgungzentrum am Evangelischen Krankenhaus Wesel GmbH, Wesel, North Rhine-Westphalia
  - Onkologie Erzgebirge, Aue-Bad Schlema, Saxony
  - Hämatologisch Onkologisches Centrum Ostsachsen ONCOS GmbH, Bautzen, Saxony
  - Fachkrankenhaus Coswig, Coswig, Saxony
  - Gemeinschaftspraxis Dr. med. Johannes Mohm Dr. med. Gabriele Prange-Krex, Dresden, Saxony
  - Gemeinschaftspraxis Hämatologie - Onkologie, Dresden, Saxony
  - Universitätsklinikum Carl Gustav Carus Dresden, Dresden, Saxony
  - Onkozentrum Dresden/Freiberg/Meißen, Dresden/Freiberg/Meißen, Saxony
  - Ambulante Onkologie Ostsachsen, Zittau, Saxony
  - Helios Klinikum Erfurt, Erfurt, Thuringia
  - Charité Universitätsmedizin Berlin, Berlin
  - Onkologische Schwerpunktpraxis Tiergarten, Berlin
  - Onkologische Schwerpunktpraxis Kurfürstendamm, Berlin
  - Praxis am Volkspark, Berlin
  - Vivantes Klinikum Neukölln, Berlin
  - Evangelische Lungenklinik Berlin, Berlin
  - DRK Kliniken Berlin Mitte, Berlin
  - Gemeinschaftskrankenhaus Havelhöhe, Berlin
  - Helios Klinikum Emil von Behring, Berlin
  - Onkologischer Schwerpunkt am Oskar-Helene-Heim, Berlin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kastner A, Kron A, Eilers L, Spier A, Mildenberger V, Simic D, Stock S, Kron F, Scheffler M, Schillinger G, van den Berg N, Wolf J, Hoffmann W. DigiNet: Optimizing personalized care for patients with stage IV non-small cell lung cancer (NSCLC) through a digitally connected provider network-analysis plan of a prospective multicenter cohort trial. J Cancer Res Clin Oncol. 2025 Sep 9;151(9):244. doi: 10.1007/s00432-025-06275-x. PMID 40924208
- See also: Project Website — https://diginet.nngm.de/